CLINICAL TRIAL: NCT05153837
Title: Effect of Oral Water in Healthy Volunteers on Cardiac Output, Regional Flow and Microcirculation in Healthy Volunteers
Acronym: WATERNAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2019_843_0064
Record Dates: First submitted 2021-11-30; First posted 2021-12-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Intravenous Fluids; Pharmacodynamics; Fluid Therapy; Fluid Responsiveness; Fluid Challenge
Keywords: intravenous fluids; pharmacodynamics; fluid therapy; fluid responsiveness; fluid challenge
MeSH Terms: interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- oral water (Experimental): Experimental group: oral administration of 500 ml of water.
  Interventions: Other: oral water
- intravenous (Active Comparator): Active comparator: Administration of 500 mL of saline (NaCl 0.9%) administered by the venous route
  Interventions: Other: saline intravenous administration

INTERVENTIONS:
Other: saline intravenous administration — Administration of 500 mL of saline (NaCl 0.9%) administered by the venous route
  Arms: intravenous
Other: oral water — 500 ml oral water
  Arms: oral water

SUMMARY:
Human digestive system physiologically ensures the absorption of oral water and hydration of the human body. Water is quickly absorbed by the digestive tract with a peak between 15 and 20 minutes. It has demonstrated that oral water remains the best hydration solution that have an effect on plasma volume expansion and cardiovascular system during exercise. While the cardiovascular effect of fluid expansion by saline serum is well known (venous return, preload and cardiac output), effect of oral water varies in the literature depending on the physiological state of the patient and the clinical state. Thus, the investigators aim to investigate oral water effects on fluid responsiveness, regional blood flow and microcirculatory changes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer subject between 18 and 30 years old
* patient with a regular sinus rhythm
* Echogenic subject.
* Fasting of solid and liquid since 8 h
* Subject in regular sinus rhythm.
* Written consent signed.

Exclusion Criteria:

* Any known cardiac, renal or endocrine pathology.
* Arrhythmia rhythm disorder by atrial fibrillation
* Pregnant or nursing woman.
* Pathology versus indicating Nacl administration.
* Person under tutors or curators or deprived of liberty.
* Person not affiliated to a social security scheme.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
number of fluid responders 30 minutes after fluid expansion | 30 minutes after fluid expansion

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens-Picardie, Amiens, France

IPD SHARING:
Plan to Share IPD: No